CLINICAL TRIAL: NCT00141297
Title: A Phase I Clinical, Pharmacokinetic, And Pharmacodynamic Evaluation Of 2 Schedules Of Oral PD 0332991, A Cyclin-Dependent Kinase Inhibitor, In Patients With Advanced Cancer
Brief Title: A Study Of Oral Palbociclib (PD-0332991), A Cyclin-Dependent Kinase Inhibitor, In Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5481001
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms; Lymphoma, Non-Hodgkin
Keywords: Advanced cancer
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD-0332991 (Experimental)
  Interventions: Drug: PD-0332991

INTERVENTIONS:
Drug: PD-0332991 — Dose ranging study - evaluating two oral schedule: (1) 3/1 Schedule - PD-0332991 administered days 1-21 of a 28-day schedule, doses ranging from 25 to 150 mg once daily; (2) 2/1 Schedule - PD-0332991 administered days 1-14 of a 21-days schedule, doses ranging from 100 to 225 mg once daily

SUMMARY:
PD-0332991 may work in cancer by stopping cancer cells from multiplying. PD-0332991 is in a new class of drugs called cyclin-dependent kinase (CDK inhibitors). This research study is the first time that PD-0332991 will be given to people. PD-0332991 is taken by mouth daily.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors (excluding SCLC and retinoblastoma) or follicular of diffuse large cell non-Hodgkin's lymphoma, histologically or cytologically proven at diagnosis which is refractory to or intolerant of established therapy know to provide clinical benefit for their condition; tumors must express Rb
* Adequate blood cell counts, kidney function and liver function and and ECOG score of 0, 1, or 2.
* Patients may have to have tumor biopsy before and after treatment.

Exclusion Criteria:

* Prior stem cell or bone marrow transplant
* Uncontrolled infection, unstable or sever intercurrent medical condition, or current drug or alcohol abuse
* Active or unstable cardiac disease or history of heart attack within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-09; Primary Completion 2008-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Abramson Cancer Center Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pharmacy/PCAM/West Pavillion, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148
- [Derived] Vaughn DJ, Flaherty K, Lal P, Gallagher M, O'Dwyer P, Wilner K, Chen I, Schwartz G. Treatment of growing teratoma syndrome. N Engl J Med. 2009 Jan 22;360(4):423-4. doi: 10.1056/NEJMc0808558. No abstract available. PMID 19164198
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481001&StudyName=A%20Study%20Of%20Oral%20Palbociclib%20%28PD-0332991%29%2C%20A%20Cyclin-Dependent%20Kinase%20Inhibitor%2C%20In%20Patients%20With%20Advanced%20Cancer%20%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- PD 0332991 25 mg QD (21/28 Days): PD 0332991 25 milligram (mg) capsule orally once daily (QD), continuously for 21 days in 28-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 50 mg QD (21/28 Days): PD 0332991 50 mg capsule orally QD, continuously for 21 days in 28-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 75 mg QD (21/28 Days): PD 0332991 75 mg capsule orally QD, continuously for 21 days in 28-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 100 mg QD (21/28 Days): PD 0332991 100 mg capsule orally QD, continuously for 21 days in 28-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 125 mg QD (21/28 Days): PD 0332991 125 mg capsule orally QD, continuously for 21 days in 28-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 150 mg QD (21/28 Days): PD 0332991 150 mg capsule orally QD, continuously for 21 days in 28-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 100 mg QD (14/21 Days): PD 0332991 100 mg capsule orally QD, continuously for 14 days in 21-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 150 mg QD (14/21 Days): PD 0332991 150 mg capsule orally QD, continuously for 14 days in 21-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 200 mg QD (14/21 Days): PD 0332991 200 mg capsule orally QD, continuously for 14 days in 21-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 225 mg QD (14/21 Days): PD 0332991 225 mg capsule orally QD, continuously for 14 days in 21-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
Period: Overall Study
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Started | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 2 | 0
Not completed — Progressive Disease | 2 | 3 | 6 | 2 | 15 | 2 | 3 | 3 | 15 | 6
Not completed — Transitioned | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all enrolled participants who received at least one dose of study medication.
Groups:
- PD 0332991 (21/28 Days): Participants received PD 0332991 capsule orally once daily (QD), continuously for 21 days in 28-day cycles in dose escalation schemes of 25 mg, 50 mg, 75 mg, 100 mg, 125 mg and 150 mg. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 (14/21 Days): Participants received PD 0332991 capsule orally once daily (QD), continuously for 14 days in 21-day cycles in dose escalation schemes of 100 mg, 150 mg and 200 mg, 225 mg. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- Total: Total of all reporting groups
Arm/Group | PD 0332991 (21/28 Days) | PD 0332991 (14/21 Days) | Total
Number analyzed (Participants) | 41 | 33 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.1) | 59.9 (11.5) | 56.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT: an adverse event occurring after initiation of PD 0332991 that met any following criteria: 1) Grade 4 hematologic toxicity (platelets less than [<] 25000 per microliter (mcL), absolute neutrophil count [ANC] <500/mcL, hemoglobin [Hb] <6.5 gram per deciliter [g/dL]; 2) ANC <1000/mcL associated with documented infection or fever greater than or equal to (>=) 38.5 degrees Celsius; 3) >=Grade 3 non-hematologic treatment-related toxicity. In an asymptomatic participant, Grade 3 corrected QT (QTc) prolongation (>500 millisecond) (only if persisted with repeat testing and after correction of reversible causes [electrolyte abnormalities or hypoxia]); and 4) Inability to receive next dose of PD 0332991 within 1 week (+/-1 day) of last dose due to lack of hematologic recovery (platelets <50000/mcL, ANC <1000/mcL, and Hb <8.0 g/dL) or due to prolonged non-hematologic toxicities of >=Grade 3 severity. Occurrence of a DLT necessitated immediate interruption of scheduled study treatment.
Time Frame: Baseline up to 28 days
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
participants | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 4 | 3

2. Primary Outcome: Maximum Administered Dose (MAD)
Description: Three new evaluable participants were to be assessed at each new dose level. The minimum time that these participants were to be followed after starting treatment was 1 cycle (28 or 21 days) before a new dose level could be opened. If none of these 3 participants experienced a DLT, the next higher dose level was to be opened on that schedule. If 1 participant developed a DLT, 3 more evaluable participants were to be enrolled at that dose level; if none of these additional 3 participants developed a DLT, the next higher dose level was to be opened on that schedule. If >=2 participants experienced a first cycle DLT at the same dose level and schedule, that dose level was to be defined as the MAD for that schedule. No additional participants were to be entered at the MAD for that dosing schedule. DLT is defined in Outcome Measure 1.
Time Frame: Baseline up to 28 days
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: milligram
Arm/Group | PD 0332991 (21/28 Days) | PD 0332991 (14/21 Days)
Number analyzed (Participants) | 41 | 33
milligram | 150 | 225

3. Primary Outcome: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose Level (RP2D)
Description: MTD was defined as the highest dose level studied for which the incidence of first cycle DLT was <33%. Once MTD was determined, it was defined as RP2D. DLT is defined in Outcome Measure 1.
Time Frame: Baseline up to 28 days
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: milligram
Arm/Group | PD 0332991 (21/28 Days) | PD 0332991 (14/21 Days)
Number analyzed (Participants) | 41 | 33
milligram | 125 | 200

4. Primary Outcome: Number of Dose-Limiting Toxicities (DLTs) Categorized as Per the Nature
Description: DLT is defined in Outcome Measure 1. Hematologic (Grade 4 [life-threatening or disabling]) and non-hematologic (Grade 3 [severe], 4 [life-threatening and disabling], 5 [resulting in death]) DLTs are reported separately. A single participant may experience more than one DLT. Both treatment-related and treatment-unrelated DLT events were reported for this outcome measure.
Time Frame: Baseline up to 28 days
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: DLTs
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
DLTs
  Hematologic DLT: Grade 4 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Non-Hematologic DLT: Grade 3 | 0 | 0 | 2 | 0 | 5 | 0 | 0 | 0 | 3 | 1
  Non-Hematologic DLT: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Non-Hematologic DLT: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events Categorized by Severity
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. For clinical description of nature (severity) of AEs, AEs were grades as: Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening or disabling AE; and Grade 5: death related to AE. AEs during Cycle 1 and AEs post Cycle 1 are reported separately.
Time Frame: Cycle 1, Cycle 2 up to 28 days after end of treatment (up to Cycle 93)
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
participants
  Cycle 1 TEAEs: Grade 1 | 0 | 2 | 1 | 0 | 7 | 1 | 2 | 2 | 6 | 1
  Cycle 1 TEAEs: Grade 2 | 1 | 1 | 2 | 1 | 5 | 0 | 0 | 1 | 6 | 1
  Cycle 1 TEAEs: Grade 3 | 0 | 0 | 3 | 2 | 7 | 1 | 0 | 0 | 8 | 2
  Cycle 1 TEAEs: Grade 4 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Cycle 1 TEAEs: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Post Cycle 1 TEAEs: Grade 1 | 0 | 0 | 1 | 0 | 8 | 0 | 0 | 1 | 3 | 1
  Post Cycle 1 TEAEs: Grade 2 | 0 | 3 | 1 | 2 | 3 | 1 | 1 | 1 | 4 | 1
  Post Cycle 1 TEAEs: Grade 3 | 2 | 0 | 2 | 0 | 3 | 2 | 1 | 1 | 8 | 3
  Post Cycle 1 TEAEs: Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Post Cycle 1 TEAEs: Grade 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Treatment-Related Treatment Emergent Adverse Events
Description: A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs during Cycle 1 and AEs post Cycle 1 are reported separately.
Time Frame: Cycle 1, Cycle 2 up to 28 days after end of treatment (up to Cycle 93)
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
participants
  Cycle 1 | 0 | 2 | 5 | 3 | 16 | 3 | 1 | 4 | 19 | 5
  Post Cycle 1 | 1 | 3 | 4 | 3 | 10 | 3 | 2 | 3 | 17 | 5

7. Primary Outcome: Number of Participants Who Died Due to Adverse Event on the Basis of Relatedness to Study Drug
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness [to study drug] was assessed by the investigator (Yes/No).
Time Frame: Baseline up to 30 days after end of treatment (up to Cycle 93)
Population: FAS included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 22 | 3 | 3 | 4 | 20 | 6
participants
  Related to Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Related to Study Drug | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1

8. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1: Single Dose
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: Pharmacokinetic (PK) analysis set included all participants from FAS who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- PD 0332991 100 mg QD: Participants who received PD 0332991 100 mg capsule orally QD, continuously for 21 days in 28-day cycles and continuously for 14 days in 21-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
- PD 0332991 150 mg QD: Participants who received PD 0332991 150 mg capsule orally QD, continuously for 21 days in 28-day cycles and continuously for 14 days in 21-day cycles. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 22 | 7 | 20 | 6
nanogram per milliliter (ng/mL) | 9.6 (6.0) | 20.7 (0.7) | 28.7 (6.9) | 45.6 (20.4) | 51.6 (22.2) | 83.8 (13.9) | 80.8 (28.4) | 104.2 (60.7)

9. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 8: Multiple Dose
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: PK analysis set included all participants from FAS who had completed PK blood sampling for at least one day. Here "N" (number of participants analyzed) signifies participant who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PD 0332991 100 mg QD: Participants who received PD 0332991 100 mg capsule orally QD, continuously for 21 days in 28-day cycles and continuously for 14 days in 21-day cycles . Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 13 | 6 | 8 | 6
ng/mL | 15.9 (5.0) | 35.7 (5.7) | 58.6 (13.9) | 71.2 (22.2) | 86.2 (29.6) | 160.8 (70.4) | 173.6 (29.5) | 185.7 (119.6)

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: The mean Cmax for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D21 for participants receiving 125 mg (21/28 Days) and Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D14 for participants receiving 200 mg (14/21 Days)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days): Participants received PD 0332991 200 mg and 125 mg capsule orally once daily (QD), continuously for 14 days in 21-day cycles and continuously for 21 days in 28-day cycles, respectively. Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
ng/mL | 104.0 (50.2)

11. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1: Food Effect
Description: To determine the impact of food (specifically a high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In this crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. The first 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, the next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results are reported as per fed and fasted conditions. The high-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of the total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 11
ng/mL
  Fed | 62.0 (20.4)
  Fasted | 44.9 (14.4)

12. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1: Single Dose
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: PK analysis set included all participants from FAS who had completed PK blood sampling for at least one day.
Measure: Median (Full Range); unit: hours
Groups:
- PD 0332991 100 mg QD: Participants who received PD 0332991 100 mg capsule orally QD, continuously for 21 days in 28-day cycles and continuously for14 days in 21-day cycles . Treatment cycles were repeated until occurrence of disease progression, unacceptable toxicity, or investigator/participant decision to withdraw from study.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 22 | 7 | 20 | 6
hours | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.3] | 4.0 [4.0 to 10.0] | 4.0 [2.0 to 10.0] | 7.0 [2.0 to 24.4] | 4.0 [4.0 to 9.8] | 5.7 [1.0 to 10.2] | 4.0 [4.0 to 7.0]

13. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 8: Multiple Dose
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 13 | 6 | 8 | 6
hours | 4.0 [2.0 to 7.0] | 4.1 [2.0 to 7.0] | 4.0 [4.0 to 9.0] | 5.5 [4.0 to 10.0] | 4.0 [1.0 to 10.0] | 7.0 [7.0 to 10.0] | 4.0 [2.0 to 7.0] | 4.5 [1.0 to 7.0]

14. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: The median Tmax for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
hours | 4.2 [2.0 to 9.8]

15. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Day 1: Food Effect
Description: To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results are reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 11
hours
  Fed | 7.00 [3.50 to 23.00]
  Fasted | 7.00 [4.00 to 10.00]

16. Primary Outcome: Terminal Half-life (t½ ) on Day 1: Single Dose
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: It was not possible to calculate data for t½ as the calculation required the slope of terminal elimination phase and the PK sampling was insufficient to characterize the terminal elimination phase, which is needed for the calculation of the t½.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Terminal Half-life (t½ ) on Day 8: Multiple Dose
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: as for outcome 16
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Terminal Half-life (t½) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half. The mean t1/2 for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
hours | 26.5 (7.0)

19. Primary Outcome: Terminal Half-life (t½ ) on Day 1: Food Effect
Description: To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 16
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

20. Primary Outcome: Area Under the Curve From Time Zero to the Last Measured Concentration (AUClast) on Day 1: Single Dose
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: PK analysis set included all participants from FAS who had completed PK blood sampling for at least one day.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hour/mL)
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 22 | 7 | 20 | 6
nanogram*hour/milliliter (ng*hour/mL) | 58 (29.5) | 134 (7.2) | 199 (40.5) | 302 (119.6) | 476 (281.1) | 594 (118.1) | 1057 (570.5) | 719 (396.7)

21. Primary Outcome: Area Under the Curve From Time Zero to the Last Measured Concentration (AUClast) on Day 8: Multiple Dose
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 13 | 6 | 8 | 6
ng*hour/mL | 118 (38.3) | 274 (41.8) | 477 (122.7) | 560 (183.1) | 722 (265.3) | 1344 (565.3) | 1395 (315.6) | 1482 (935.1)

22. Primary Outcome: Area Under the Curve From Time Zero to the Last Measured Concentration (AUClast) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). The mean AUClast for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
ng*hour/mL | 3626 (2565.8)

23. Primary Outcome: Area Under the Curve From Time Zero to the Last Measured Concentration (AUClast) on Day 1: Food Effect
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results are reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 11
ng*hour/mL
  Fed | 809 (372.7)
  Fasted | 668 (280.6)

24. Primary Outcome: Area Under the Curve From Time Zero to End of the Dosing Interval [AUC(0 to Tau)] on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Area under the curve from time zero to end of the dosing interval (24 hours) [AUC (0-tau)]. The mean AUC (0-tau) for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
ng*hour/mL | 1863 (1096.5)

25. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] on Day 1: Single Dose
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: It was not possible to calculate data for this outcome measure because calculation was dependent on the linear regression of data points collected during the terminal phase and the PK sampling was insufficient to characterize the terminal phase, which is needed for the calculation of the AUC (0 - ∞).
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] on Day 8: Multiple Dose
Description: as for outcome 25
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: as for outcome 25
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] on Day 1: Food Effect
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 25
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

28. Primary Outcome: Apparent Oral Clearance (CL/F) on Day 1: Single Dose
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: It was not possible to calculate data for this outcome measure because calculation was dependent on the linear regression of data points collected during the terminal phase and the PK sampling was insufficient to characterize the terminal phase, which is needed for the calculation of the CL/F.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Apparent Oral Clearance (CL/F) on Day 8: Multiple Dose
Description: as for outcome 28
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: as for outcome 28
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: Apparent Oral Clearance (CL/F) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Clearance of a drug is a measure of rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. The mean CL/F for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
liter/hour | 86.1 (42.8)

31. Primary Outcome: Apparent Oral Clearance (CL/F) on Day 1: Food Effect
Description: Clearance of a drug is a measure of rate at which a drug is metabolized or eliminated by normal biological processes. To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 28
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

32. Primary Outcome: Apparent Volume of Distribution (Vz/F) on Day 1: Single Dose
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: It was not possible to calculate data for this outcome measure because calculation was dependent on the linear regression of data points collected during the terminal phase and the PK sampling was insufficient to characterize the terminal phase, which is needed for the calculation of the Vz/F.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

33. Primary Outcome: Apparent Volume of Distribution (Vz/F) on Day 8: Multiple Dose
Description: as for outcome 32
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: as for outcome 32
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Primary Outcome: Apparent Volume of Distribution (Vz/F) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed. The mean Vz/F for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
liter | 3103 (1237.8)

35. Primary Outcome: Apparent Volume of Distribution (Vz/F) on Day 1: Food Effect
Description: Volume of distribution: theoretical volume in which total amount of drug would need to be uniformly distributed to produce desired plasma concentration. To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 32
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

36. Primary Outcome: Accumulation Ratio (Rac) on Day 8: Multiple Dose
Description: Rac at Day 8 = AUC (0-tau) at Day 8 divided by AUC (0-tau) at Day 1.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10, and 24 hours post-dose on C1D1 and C1D8
Population: It was not possible to calculate data for this outcome measure because calculation was dependent on the linear regression of data points collected during the terminal phase and the PK sampling was insufficient to characterize the terminal phase, which is needed for the calculation of the Rac.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Primary Outcome: Accumulation Ratio (Rac) on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Rac at Day 14/21 = AUC (0-tau) at Day 14/21 divided by AUC (0-tau) at Day 1. The mean Rac for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
ratio | 2.5 (0.8)

38. Primary Outcome: Terminal Phase Rate Constant [Lambda (z)] on Day 1: Single Dose
Description: Terminal phase rate constant is the absolute value of the slope of a linear regression during the terminal phase of the natural--logarithm transformed concentration--time profile.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 1 of Cycle 1 (C1D1)
Population: It was not possible to calculate data as the calculation required the slope of terminal elimination phase and the PK sampling was insufficient to characterize the terminal elimination phase
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Primary Outcome: Terminal Phase Rate Constant [Lambda (z)] on Day 8: Multiple Dose
Description: Terminal phase rate constant is the absolute value of the slope of a linear regression during the terminal phase of the natural-logarithm transformed concentration-time profile.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, and 10 hours post-dose on Day 8 of Cycle 1 (C1D8)
Population: It was not possible to calculate the data as the calculation required the slope of terminal elimination phase and the PK sampling was insufficient to characterize the terminal elimination phase.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Primary Outcome: Terminal Phase Rate Constant [Lambda (z)] on Day 14/21 Dose-Corrected to 125 mg: Multiple Dose
Description: Terminal phase rate constant is the absolute value of the slope of a linear regression during the terminal phase of the natural-logarithm transformed concentration-time profile. The mean lambda (z) for 200 mg dose group (dose corrected to 125 mg) on Cycle 1 Day 14 (C1D14) and 125 mg dose group on Cycle 1 Day 21 (C1D21) was calculated. Only participants from 125 mg and 200 mg dose groups were reported.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 13
1/hour | 0.028 (0.0)

41. Primary Outcome: Terminal Phase Rate Constant [Lambda (z)] on Day 1: Food Effect
Description: Terminal phase rate constant: absolute value of slope of a linear regression during terminal phase of natural-logarithm transformed concentration-time profile. To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose), 1, 2, 4, 7, 10 and 24 hours post-dose on C1D1, C2D1
Population: as for outcome 39
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

42. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in the Urine (Ae): Single Dose
Description: Ae is the cumulative amount of drug recovered unchanged in urine over the 10 hour collection interval. Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval. Urine PK analysis was performed only in the MTD/RP2D groups (125 mg [21/28 Days] and 200 mg [14/21 Days]).
Time Frame: Hour 0 (pre-dose) to 10 hours post-dose on C1D1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 200 mg QD (14/21 Days)
Number analyzed (Participants) | 9 | 10
microgram (mcg) | 2191 (1404) | 3171 (2442)

43. Primary Outcome: Cumulative Amount of Drug Recovered Unchanged in the Urine (Ae): Food Effect
Description: The Ae is defined in Outcome Measure 42. To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose) to 10 hours post-dose on C1D1
Population: Data was not collected because urine PK was not planned to be analyzed by food effect, as per protocol.
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

44. Primary Outcome: Percent Dose Recovered Unchanged in Urine (Percent Ae): Single Dose
Description: Percent of dose recovered unchanged in urine over the 10 hour collection interval=100*(Ae divided by dose). Ae is the cumulative amount of drug recovered unchanged in urine over the 10 hour collection interval. Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval.
Time Frame: Hour 0 (pre-dose) to 10 hours post-dose on C1D1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 200 mg QD (14/21 Days)
Number analyzed (Participants) | 9 | 10
percentage of dose | 1.75 (1.1) | 1.59 (1.2)

45. Primary Outcome: Percent Dose Recovered Unchanged (Percent Ae) in Urine: Food Effect
Description: The percent Ae is defined in Outcome Measure 44. To determine impact of food (specifically high-fat meal) on PD 0332991 PK, participants were tested under fed and fasted conditions in crossover fashion. Each participant served as their own control. In crossover fashion first dose was administered under either fed (high-fat meal) or fasted (10-hour fast) condition on Day 1 of Cycle 1 and 2. First 6 participants were tested under fed (on C1D1) followed by fasted (on C2D1) conditions, next 6 participants were tested under fasted (on C1D1) followed by fed (on C2D1) conditions. Only participants in PD 0332991 200 mg (14/21 days) and 125 mg (21/28 days) groups participated in food effect crossover and results were to be reported as per fed and fasted conditions. High-fat meal was composed of around 800 to 1000 calories total, with fat composing around 50% of total caloric content.
Time Frame: Hour 0 (pre-dose) to 10 hours post-dose on C1D1
Population: Data was not collected because urine PK was not planned to be analyzed by food effect, as per protocol.
Arm/Group | PD 0332991 200 mg (14/21 Days) and 125 mg (21/28 Days)
Number analyzed (Participants) | 0

46. Primary Outcome: Number of Participants With Best Response
Description: Number of participants with best response. Complete response (CR): disappearance of all target and non-target lesions. Partial Response (PR): >=30% decrease in sum of longest diameter (LD) of lesions taking as reference baseline sum LD and no unequivocal progression in non-target lesions. Progressive disease (PD): >=20% increase in sum of LD of lesions taking as a reference smallest sum of the LD since treatment start, or the appearance of >=1 new lesion or unequivocal progression of existing non-target lesions. Stable disease (SD): neither shrinkage for PR nor increase for PD taking as reference smallest sum of LD since treatment start. SD was assessed following the first 2 cycles of treatment (>=2 cycles), 4 cycles of treatment (>=4 cycles), and 10 cycles of treatment (>=10 cycles). Participants may be reported in more than 1 category of SD. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response.
Time Frame: Baseline up to end of treatment, assessed at C1D1, C1D8, C1D15, C1D22, thereafter Day 1, 8, 15, and 22 of every other cycle up to end of treatment (up to Cycle 93)
Population: Modified Full Analysis Set included all enrolled participants who received at least 1 dose of study medication in Cycle 1 and completed a post-treatment response assessment.
Measure: Number; unit: participants
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 20 | 2 | 3 | 3 | 19 | 6
participants
  Confirmed CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confirmed PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  SD >=2 Cycles | 1 | 2 | 1 | 1 | 6 | 2 | 1 | 0 | 5 | 3
  SD >=4 Cycles | 1 | 2 | 1 | 1 | 3 | 2 | 1 | 0 | 3 | 2
  SD >=10 Cycles | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1
  PD | 2 | 1 | 6 | 2 | 13 | 0 | 2 | 3 | 12 | 3
  Not Assessable | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

47. Primary Outcome: Inhibition of Cyclin-dependent Kinases 4 and 6 (Cdk4/6) Based on Phosphorylated Retinoblastoma (p-Rb) in Tumor Tissue
Description: Phosphorylation of the retinoblastoma (Rb) protein by Cdk4/6 is typically required for human cancer cell proliferation. Tumor biopsies were to be performed, to demonstrate inhibition of Cdk4/6 based on reduction in phosphorylated Rb (p-Rb) in tumor tissue and p-Rb levels (fold decrease) were to be reported.
Time Frame: Baseline, C1D1, C1D8, C1D15, C1D22, thereafter Day 1, 8, 15, and 22 of every other cycle up to end of treatment (up to Cycle 93)
Population: Data was reported in individual participant listings and not summarized due to change in planned analysis, where baseline and post-baseline tumor biopsies for biomarkers were no longer required and were not obtained for all participants.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

48. Primary Outcome: Correlation of Cyclin-dependent Kinases 4 and 6 (Cdk4/6) With PD 0322991 Dose
Description: Phosphorylation of the retinoblastoma (Rb) protein by Cdk4/6 is typically required for human cancer cell proliferation. Tumor biopsies were to be performed, to demonstrate inhibition of Cdk4/6 based on reduction in phosphorylated Rb (p-Rb) in tumor tissue, in correlation with respect to PD 0322991 dose.
Time Frame: as for outcome 47
Population: as for outcome 47
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Primary Outcome: Correlation of Cyclin-dependent Kinases 4 and 6 (Cdk4/6) With Exposure
Description: Phosphorylation of the retinoblastoma (Rb) protein by Cdk4/6 is typically required for human cancer cell proliferation. Tumor biopsies were to be performed, to demonstrate inhibition of Cdk4/6 based on reduction in phosphorylated Rb (p-Rb) in tumor tissue, in correlation with PD 0322991 exposure.
Time Frame: as for outcome 47
Population: as for outcome 47
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Primary Outcome: Correlation of Cyclin-dependent Kinases 4 and 6 (Cdk4/6) With Tumor Response
Description: Phosphorylation of the retinoblastoma (Rb) protein by Cdk4/6 is typically required for human cancer cell proliferation. Tumor biopsies were to be performed, to demonstrate inhibition of Cdk4/6 based on reduction in phosphorylated Rb (p-Rb) in tumor tissue, in correlation with tumor response.
Time Frame: as for outcome 47
Population: as for outcome 47
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PD 0332991 25 mg QD (21/28 Days) | PD 0332991 50 mg QD (21/28 Days) | PD 0332991 75 mg QD (21/28 Days) | PD 0332991 100 mg QD (21/28 Days) | PD 0332991 125 mg QD (21/28 Days) | PD 0332991 150 mg QD (21/28 Days) | PD 0332991 100 mg QD (14/21 Days) | PD 0332991 150 mg QD (14/21 Days) | PD 0332991 200 mg QD (14/21 Days) | PD 0332991 225 mg QD (14/21 Days)
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 3/7 | 1/3 | 3/22 | 0/3 | 2/3 | 3/4 | 4/20 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 3/3 | 22/22 | 3/3 | 3/3 | 4/4 | 20/20 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD 0332991 25 mg QD (21/28 Days) (N=3) | PD 0332991 50 mg QD (21/28 Days) (N=3) | PD 0332991 75 mg QD (21/28 Days) (N=7) | PD 0332991 100 mg QD (21/28 Days) (N=3) | PD 0332991 125 mg QD (21/28 Days) (N=22) | PD 0332991 150 mg QD (21/28 Days) (N=3) | PD 0332991 100 mg QD (14/21 Days) (N=3) | PD 0332991 150 mg QD (14/21 Days) (N=4) | PD 0332991 200 mg QD (14/21 Days) (N=20) | PD 0332991 225 mg QD (14/21 Days) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stent placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD 0332991 25 mg QD (21/28 Days) (N=3) | PD 0332991 50 mg QD (21/28 Days) (N=3) | PD 0332991 75 mg QD (21/28 Days) (N=7) | PD 0332991 100 mg QD (21/28 Days) (N=3) | PD 0332991 125 mg QD (21/28 Days) (N=22) | PD 0332991 150 mg QD (21/28 Days) (N=3) | PD 0332991 100 mg QD (14/21 Days) (N=3) | PD 0332991 150 mg QD (14/21 Days) (N=4) | PD 0332991 200 mg QD (14/21 Days) (N=20) | PD 0332991 225 mg QD (14/21 Days) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1 | 6 | 1 | 1 | 1 | 8 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 3 | 8 | 3 | 0 | 0 | 12 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 5 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Middle ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 4 | 0 | 0 | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 5 | 0 | 2 | 2 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 4 | 0 | 2 | 1 | 9 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 3 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 6 | 2 | 1 | 1 | 11 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 6 | 1 | 1 | 1 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 3 | 2 | 10 | 3 | 2 | 1 | 15 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 4 | 0
Pain (General disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 4 | 0
Peripheral coldness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Ulcer (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver palpable subcostal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Waist circumference increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 1 | 3 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 4 | 1 | 1 | 0 | 4 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Onychomalacia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cast application (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.